CLINICAL TRIAL: NCT06859632
Title: Effect on Healthcare Professionals' Self-efficacy of a 45-minute vs Three-hour Educational Intervention on Communication and Play in Paediatric Clinical Practice: A Randomised Controlled Trial Study Protocol
Brief Title: 45 Minutes Vs. Three Hours Educational Intervention on Communication and Play for Paediatric Healthcare Professionals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jakob Thestrup Hansen, MscGH, PhD candidate, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P-2021-426
Record Dates: First submitted 2025-02-25; First posted 2025-03-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Education; Communication; Play; Pediatrics
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 45-minute educational intervention (Active Comparator): Participants will receive a 45-minute educational intervention on communication and the use of play in paediatric clinical practice
  Interventions: Other: 45-minute educational intervention
- 3-hour educational intervention (Experimental): Participants will receive a 3-hour educational intervention on communication and the use of play in paediatric clinical practice
  Interventions: Other: 3-hour educational intervention

INTERVENTIONS:
Other: 3-hour educational intervention — A 3-hour educational intervention on communication and the use of play in paediatric clinical practice.
  Participants in both arms will have access to written learning material and an app that has been developed.
  Arms: 3-hour educational intervention
Other: 45-minute educational intervention — A 45-minute educational intervention on communication and the use of play in paediatric clinical practice.
  Participants in both arms will have access to written learning material and an app that has been developed.
  Arms: 45-minute educational intervention

SUMMARY:
The goal for this trial is to test the effect of an educational programme on communication and play for healthcare professionals working with children and adolescents. The main questions to answer are:

1. Does a 45-minute educational intervention on communication and play have the same effect on healthcare professionals' self-efficacy in patient-centredness compared with a three-hour intervention?
2. What is the effect of the intervention on participants' motivation to engage in the educational activity, cognitive load, knowledge, satisfaction, and the impact on their individual practice ?

Participants will be randomly assigned to either a 45-minute or a three-hour educational intervention. They will complete a questionnaire at three time points: before the intervention, immediately after, and at a 12-week follow-up.

DETAILED DESCRIPTION:
BACKGROUND: Communication is an essential skill for all healthcare professionals working with children and adolescents in hospitals. There is growing focus on child-centred communication, which emphasize communicating directly with children and adolescents in healthcare rather than focusing on the parents. However, educational programmes for this remain limited while those that exist are heterogenous and often assessed without comparison groups or validated tools.

OBJECTIVE: To investigate the effect on healthcare professionals' self-efficacy of a 45-minute vs three-hour educational intervention on communication and the use of play in clinical paediatric practice

INTERVENTION: This trial evaluates the educational programme "Communication and Play with Children and Adolescents in Healthcare", which focuses on age-appropriate communication with paediatric patients, including the deliberate use of play. The trial compares two educational interventions that differ in duration (45 minutes vs. three hours) and learning methods. While both interventions include didactic learning, reflection, and discussions, the three-hour session adds role-play activities, whereas the 45-minute session delivers a condensed version without role-play.

DESIGN: Single-centre, randomized, controlled, two-arm, noninferiority trial. A noninferiority design is used to assess whether there is a difference between the two educational interventions or if the 45-minute educational intervention is comparable to the three-hour educational intervention.

SETTING: The University Hospital of Copenhagen - Rigshospitalet, Denmark.

RECRUITMENT: All healthcare professionals working in the Department of Paediatrics and Adolescent Medicine at Rigshospitalet will be eligible to participate. Potential participants will be contacted by their leaders and be informed of the study. A written consent will then be obtained.

SAMPLE SIZE: The sample size calculation assumes that the 45-minute intervention is as effective as the three-hour intervention for the primary outcome (self-efficacy). A non-inferiority margin of 0.25 points is set, meaning the mean self-efficacy score for the 45-minute intervention can be up to 0.25 points lower than that of the three-hour intervention without being considered inferior. Based on a one-sided two-sample t-test with a margin of 0.25, an alpha of 0.025, a power of 80%, and a standard deviation of 0.45 derived from the pilot study, the required sample size is 52 participants per group. Since the intervention is conducted in clusters of 25 participants, the sample size calculation is adjusted for cluster randomization by multiplying by the design effect, calculated as 1 + (cluster size - 1) × ICC. Assuming an ICC of 0.01 results in a design effect of 1.24 and an adjusted sample size of 65 per group. Accounting for a 10% dropout rate, the final required sample size is 72 per group. It is planned to include a total of 150 participants.

RANDOMIZATION: Eligible participants will be randomly assigned in a 1:1 ratio to either a 45-minute educational intervention or a three-hour educational intervention using computer-generated block randomization through REDCap. The randomization process will ensure an interprofessional distribution of participants in each intervention group. Both the statistician and the researchers conducting the analysis will be blinded to participant allocation.

ETHICS: This trial complies with the principles outlined in the Declaration of Helsinki for biomedical research. Approval has been obtained from the Danish Data Protection Agency (P-2021-426). The study was approved but deemed exempt from requiring ethical approval by The Scientific Ethical Committees for the Capital Region of Denmark (Journal-nr.: H-21028050). Participation is entirely voluntary, and both educational interventions will take place during working hours at no cost to the participants. Participants may withdraw from the study at any time without any repercussions. To ensure confidentiality, all data will be securely stored in a protected database.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals employed in the Department of Paediatrics and Adolescent Medicine at Rigshospitalet (nurses, doctors, physiotherapist, occupational therapists, dieticians, medical secretaries, and social workers)
* Provide signed informed consent before randomisation

Exclusion Criteria:

* Staff taking part in planning of the intervention
* Lack of informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | From enrollment to 12-week follow-up
  Self-efficacy measured using a 10-item questionnaire on a 5-point likert scale (1 = very low degree, 5 = very high degree). Questions are adapted from the Danish version of the validated Self-Efficacy in Patient-Centeredness Questionnaire (SEPCQ-27).This questionnaire evaluates participants' confidence in their ability to build relationships and communicate with children and adolescents in hospital settings.

SECONDARY OUTCOMES:
Motivation | Immediately after intervention
  Motivation measured by using the validated Intrinsic Motivation Inventory (IMI). The IMI is a self-report questionnaire that measures a person's subjective experience related to a specific activity on a Likert scale ranging from 1 (Not at all true) to 7 (Very true). The standard IMI includes 22 items. For this study, the 7-item Interest/Enjoyment subscale is used, which is considered to directly measure intrinsic motivation related to a recently completed activity.
Self-evaluated knowledge about paediatric communication | From enrollment to 12 week follow-up
  The participants self-perceived knowledge about paediatric communication will be assessed using a single item. The question is "What is your knowledge about age-appropriate communication with children and adolescents?" (5 point Likert scale from "no knowledge" to "very high knowledge").
Cognitive load | Immediately after intervention
  Measured using the Mental effort rating scale by Paas (1992). This validated, single item measure asks participants to rate their perceived mental effort ranging from "very, very low mental effort" to "very, very high mental effort" on a 9-point Likert scale.
Satisfaction with intervention | Immediately after intervention
  Participant satisfaction will be measured using a pre-designed questionnaire to assess participants' perceptions and satisfaction with the interventions. It will include five items covering relevance to clinical practice, overall quality, and whether they would recommend it to other healthcare professionals. One open-ended questions will invite participants to share general feedback and any additional comments about their experience.
Impact on individual practice and training need | 12 week follow-up
  Impact on individual practice and training needs will be evaluated through five items that examine whether participants changed their own practice, engaged with further reading, or identified a need for more training. Possible scores range from 1 (not at all) to 5 (to a very high degree).

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data to replicate the analysis will be available from the corresponding author (ORCID: 0000-0002-0093-8555) on reasonable request until five years after completion of the study, according to Danish law.

REFERENCES:
- [Background] Krebs CL, Thestrup J, Hybschmann J, Graber K, Gjaerde LK, Topperzer MK, Nielsen ET, Larsen A, Ramchandani P, Frandsen TL, Sorensen JL. A BEME review of educational programmes on the use of play in paediatric practice: BEME Guide No. 82. Med Teach. 2024 Nov;46(11):1393-1403. doi: 10.1080/0142159X.2023.2287983. Epub 2023 Dec 14. PMID 38098168
- [Background] Thestrup J, Sorensen JL, Esbjorn BH, Hybschmann J, Frandsen TL, DeCosta P, Gjaerde LK. Paediatric patient perceptions of healthcare professionals: contributions to a communication curriculum. Eur J Pediatr. 2024 Dec 12;184(1):75. doi: 10.1007/s00431-024-05911-x. PMID 39663230
- [Background] Jeppesen E, Schmidt AA, Skjodt CK, Hybschmann J, Gjaerde LK, Thestrup J, Hansson H, Sorensen JL. Educational programmes for paediatric healthcare professionals in patient- and family-centred care. A scoping review. Eur J Pediatr. 2024 May;183(5):2015-2028. doi: 10.1007/s00431-024-05455-0. Epub 2024 Mar 2. PMID 38430279
- [Background] Thestrup J, Sorensen JL, Hybschmann J, Topperzer MK, Graber K, O'Farrelly C, Gibson J, Ramchandani P, Frandsen TL, Gjaerde LK. Establishing consensus on principles and competencies for the use of play in clinical practice in hospitals: An international Delphi study. Eur J Pediatr. 2024 Apr;183(4):1595-1605. doi: 10.1007/s00431-023-05411-4. Epub 2024 Jan 6. PMID 38183437
- [Background] Gjaerde LK, Hybschmann J, Dybdal D, Topperzer MK, Schroder MA, Gibson JL, Ramchandani P, Ginsberg EI, Ottesen B, Frandsen TL, Sorensen JL. Play interventions for paediatric patients in hospital: a scoping review. BMJ Open. 2021 Jul 26;11(7):e051957. doi: 10.1136/bmjopen-2021-051957. PMID 34312210
- [Background] Davison G, Conn R, Kelly MA, Thompson A, Dornan T. Fifteen-minute consultation: Guide to communicating with children and young people. Arch Dis Child Educ Pract Ed. 2023 Apr;108(2):91-95. doi: 10.1136/archdischild-2021-323302. Epub 2021 Dec 2. PMID 34857651
- [Background] Hoeg BL, Sevillano PB, Enesco I, Wakefield CE, Larsen HB, Bidstrup PE. Child-centered communication interventions in pediatric oncology: A scoping review and proposed new communication model. Pediatr Blood Cancer. 2023 Jul 4:e30533. doi: 10.1002/pbc.30533. Online ahead of print. PMID 37401446
- [Derived] Thestrup J, Sorensen JL, Bidstrup PE, Rosthoj S, Hybschmann J, Esbjorn BH, Dybdal D, Barslund K, Topperzer MK, Frandsen TL, Gjaerde LK. Effect on healthcare professionals' self-efficacy of a 45-min versus 3-hour educational intervention on communication and play in paediatric clinical practice in Denmark: a randomised controlled trial study protocol. BMJ Open. 2025 Sep 14;15(9):e101703. doi: 10.1136/bmjopen-2025-101703. PMID 40953883